CLINICAL TRIAL: NCT01440426
Title: Connective Tissue Graft vs Mucograft Collagen Matrix for Coverage of Multiple Gingival Recession Defects Randomized Controlled Clinical Trial Assessing Superiority in Health Related Quality of Life and Non-Inferiority in Root Coverage
Brief Title: Connective Tissue Graft Versus Mucograft Collagen Matrix for Coverage of Multiple Gingival Recession Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maurizio Tonetti (Network)
Collaborators: The European Research Group on Periodontology (ERGOPerio) (Network)
Responsible Party: Sponsor-Investigator, Maurizio Tonetti, Executive DIrector, The European Research Group on Periodontology (ERGOPerio)
Organization: The European Research Group on Periodontology (ERGOPerio) (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERGOPerio 11-01
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Gingival Recession
Keywords: gingival recession; root coverage; periodontal surgery; collagen matrix; mucograft; multiple exposed teeth
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous connective tissue graft (Active Comparator): Soft tissue harvested from patient palate
  Interventions: Procedure: Autologous connective tissue graft with rotated papilla flap
- Collagen Matrix Construct (Experimental): Mucograft collagen matrix manufactured by Geistlich AG, Switzerland
  Interventions: Device: Collagen matrix construct (Mucograft)

INTERVENTIONS:
Procedure: Autologous connective tissue graft with rotated papilla flap — Subepithelial connective tissue graft harvested from hard palate
  Other Names: Subepithelial connective tissue graft
  Arms: Autologous connective tissue graft
Device: Collagen matrix construct (Mucograft) — Mucograft Collagen Matrix combined with rotated papilla flap
  Other Names: Mucograft gingival augmentation
  Arms: Collagen Matrix Construct

SUMMARY:
This study deals with coverage of multiple denuded roots. The current standard treatment requires surgical correction and uses soft tissue taken from the roof of the mouth to enhance results. The hypothesis of this trial is that a synthetic collagen matrix (called Mucograft) can be used to replace soft tissue taken from the subject. If the collagen matrix will prove to be equally as effective as the patient own tissue, it will be possible to avoid a more extensive surgery and decrease pain and discomfort.

DETAILED DESCRIPTION:
Objectives The main objective of this study is to assess if the Mucograft Collagen Matrix reduces morbidity, shortens time to recovery and improves patient based outcomes with respect to the use of autologous connective tissue graft harvested from the patient own palate when used to obtain root coverage of multiple adjacent gingival recessions.

The secondary objective is to assess the non-inferiority - in terms of complete root coverage, percentage of root coverage and professional evaluation of aesthetics - of the use of Mucograft Collagen Matrix and autologous connective tissue harvested from the patient's own palate.

Design and Outcomes This will be a parallel group, standard of care-controlled, assessor-blind, randomized, multicenter, multinational, clinical trial.

The statistical design will be a superiority trial in terms of the primary outcomes (patient based outcomes) and non-inferiority trial in terms of the professional outcomes measuring root coverage and aesthetics.

Sample size has been estimated in 140 subjects per treatment arm using a pilot case series analyzed with a multilevel statistical approach and a non inferiority margin of 0.25 mm in recession coverage.

Randomization will be performed by computer generated random codes, using random permuted blocks with a block size of 4 to avoid uneven splits and minimization for the key prognostic factor cigarette smoking. Allocation will be concealed to the surgeons until completion of preparation of the recipient bed by opaque envelopes. A central study registrar will perform patient registration.

Study locations will include academic centers and a practice-based research network in Italy, Switzerland, Germany, Belgium, France, Spain and Greece.

A single examiner, blind with respect to the treatment assignment, will perform all measurements at each center. Trained personnel not involved with the surgical intervention will: i) administer patient questionnaires, ii) provide instructions and collect patient diaries. A single calibrated investigator with specific experience in using the specific score will centrally perform assessment of esthetic scores on standardized digital images.

A biostatistician blind with respect to treatment assignment will perform the analysis.

Interventions and Duration The two intervention groups will consist of surgery with connective tissue graft (standard of care control) and surgery with the application of Mucograft Collagen Matrix (MCM, Test group). Experienced clinicians will deliver treatment consisting of root coverage surgery using coronally advanced flaps, the most utilized procedure for coverage of multiple recessions. Surgery will be standardized and the same procedures/materials will be employed to ensure consistency.

Follow-up of individual patients will be 6 months (to be extended to 3 years if funding will be available)

ELIGIBILITY:
Inclusion Criteria:

* 2-4 adjacent gingival recession (one at least 3 mm deep)

Exclusion Criteria:

* Interdental attachment loss greater than 1 mm at recession sites

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Time to recovery after surgery | 3 months
  Time to recover after surgery assessed by diary and post'op follow up professional assessment

SECONDARY OUTCOMES:
Complete root coverage | 6 months
  Frequency of complete root coverage
Percentage of root coverage | 6 months
  Percentage of the exposed tooth root covered after surgical intervention
Esthetics | 6 months
  Professional assessment by blind assessor of the esthetic result

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD PhD, Principal Investigator — The European Research Group on Periodontology (ERGOPerio); Pierpaolo COrtellini, MD, Principal Investigator — The European Research Group on Periodontology (ERGOPerio)
Locations (13):
- ICPDOI, Brussels, Belgium
- Germany (4):
  - Praxis Dr. Halben, Hamburg
  - Praxis Prof Huerzeler - Dr Zuhr, Munich
  - Praxis Prof Wachtel - Dr Bolz, Munich
  - Praxis Prof. Topoll, Münster
- Clinic Fourmousis, Athens, Greece
- Italy (3):
  - University of FLorence, Florence
  - Practice Prof Giulio Rasperini, Piacenza
  - University of Pisa, Pisa
- Spain (2):
  - Clinia Zabalegui, Bilbao
  - Clinica Guerrero, Málaga
- Switzerland (2):
  - Praxis Wallkamm, Langenthal
  - Praxis Burkhardt, Zurich